CLINICAL TRIAL: NCT03986554
Title: Swallowing Pressure Profiles in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB201901651; OCR24403 (Other: UF OnCore)
Record Dates: First submitted 2019-06-13; First posted 2019-06-14 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Healthy
Keywords: Swallowing

STUDY DESIGN:
Intervention Model Description: Participants will include healthy adults, between the ages of 18 and 45 years with no major medical history.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomization Visit A (Other): Participants enrolled in this arm will consume 300ml of water over 60 minutes. Each session will consist of 30 swallows broken into three 10-swallow sequences of 10ml of water. Each sequence will be use VFSS to visualize swallows.
  Interventions: Procedure: Videofluoroscopic swallow study
- Randomization Visit B (Other): Participants enrolled in this arm will consume 300ml of water over 60 minutes. Each session will consist of 30 swallows broken into three 10-swallow sequences of 10ml of water. Sequences 1 and 3 will use videofluoroscopy only, while sequence 2 will use VFSS with simultaneous pharyngeal high resolution manometry in order to visualize swallows.
  Interventions: Procedure: Videofluoroscopic swallow study; Procedure: pharyngeal High Resolution Manometry

INTERVENTIONS:
Procedure: Videofluoroscopic swallow study — The Swallowing Systems Core laboratory is fully equipped to perform VFSS with a C-arm (OEC 9900) that is dedicated solely for research purposes. VFSS recordings will be kept to a minimum and only turned on during the execution of each swallow in all sequences. Video recording and images captured during the VFSS will be synced and saved to a secure server for data analysis. VFSS allows for time-synced, frame-by-frame data analysis for the specific measures taken during swallowing tasks. The physiological swallowing measures (temporal and kinematic movement of the hyolaryngeal complex during swallowing) cannot be visualized with any other technique. Patients will swallow only water. Aspiration (bolus into trachea) is not expected to occur during this study given that the individuals recruited will have no prior history of disease or disorder, and aspiration is uncommon in healthy individuals.
  Other Names: VFSS, x-ray of swallowing
Procedure: pharyngeal High Resolution Manometry — This procedure will only take place once during sequence 2 of the randomization B session. If desired, a small amount (< 0.5 mL) of topical 2% viscous lidocaine hydrochloride will be applied to the participant's nostril of choice prior to catheter insertion. The catheter will be placed through the nasal passage, oropharynx, and hypopharynx to the esophagus. Correct catheter placement will be verified with VFSS. With the catheter in place, the subject will perform 10 swallows of 10ml and is expected to take approximately 2.5 minutes. The catheter will then be removed and the subject will move on to sequence 3. Individuals have the option to decline this procedure if it is uncomfortable or difficult to tolerate.
  Other Names: pHRM, HRM
  Arms: Randomization Visit B

SUMMARY:
This study is designed to determine the impact of a pharyngeal High Resolution Manometry catheter on swallowing biomechanics

DETAILED DESCRIPTION:
During pharyngeal High Resolution Manometry (pHRM) a small bore flexible catheter is introduced into the pharynx to detect intrabolus pressure and contact of pharyngeal structures during swallowing. The presence of the catheter through the upper esophageal sphincter (UES) leads to a violation of its natural closed state. It is not clear how this intrusion influences the swallowing biomechanics . Hence, this project's goal is to identify how hyoid movement is altered during swallowing with the presence of a pHRM catheter in place.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults between the ages of 18-45 with no major medical conditions.
* no specific gender or race will be excluded or targeted for participation in this study.

Exclusion Criteria:

* adults who are pregnant
* adults with swallowing impairment, brain injury, deviated septum, G.I. strictures, obstructions, or Zenker's diverticulum, surgeries to nose, neck, or throat, or bleeding disorders will be excluded from this study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Change in peak anterior and superior hyoid movement | Baseline; Week 1
  peak hyoid movement (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Emily K Plowman, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No